CLINICAL TRIAL: NCT05478863
Title: A Double-Blind, Randomized, Placebo-Controlled, Within-Subject Crossover Study of the Effects of Combinations of Cannabinoids and Caffeine
Brief Title: The Pharmacodynamics of Cannabinoid-Caffeine Combinations
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Canopy Growth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00330923
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Behavioral Pharmacology of Cannabinoids
MeSH Terms: interventions — Dronabinol; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Oral placebo (Placebo Comparator): Acute administration of oral placebo three times in study session (Time 0, 60, and 120).
  Interventions: Drug: Oral Placebo
- Oral administration of 2.5 mg THC (Experimental): Acute administration of oral THC (2.5 mg) three times in study session (Time 0, 60, and 120).
  Interventions: Drug: Oral THC
- Oral administration of 2.5 mg THC + 60 mg caffeine (Experimental): Acute administration of oral THC (2.5 mg) and oral caffeine (60 mg) three times in study session (Time 0, 60, and 120).
  Interventions: Drug: Oral THC; Drug: Oral Caffeine
- Oral administration of 2.5 mg THC + 60 mg caffeine + 35 mg CBD (Experimental): Acute administration of oral THC (2.5 mg), oral caffeine (60 mg), and oral CBD (35 mg) three times in study session (Time 0, 60, and 120).
  Interventions: Drug: Oral THC; Drug: Oral CBD; Drug: Oral Caffeine

INTERVENTIONS:
Drug: Oral Placebo — Placebo will be orally self-administered by study participants.
  Arms: Oral placebo
Drug: Oral THC — THC will be orally self-administered by study participants.
  Arms: Oral administration of 2.5 mg THC; Oral administration of 2.5 mg THC + 60 mg caffeine; Oral administration of 2.5 mg THC + 60 mg caffeine + 35 mg CBD
Drug: Oral CBD — CBD will be orally self-administered by study participants.
  Arms: Oral administration of 2.5 mg THC + 60 mg caffeine + 35 mg CBD
Drug: Oral Caffeine — Caffeine will be orally self-administered by study participants.
  Arms: Oral administration of 2.5 mg THC + 60 mg caffeine; Oral administration of 2.5 mg THC + 60 mg caffeine + 35 mg CBD

SUMMARY:
Cannabis and caffeine are two of the most commonly consumed psychoactive substances in the world, with many consumers reporting positive impacts on energy, alertness, and focus. Preliminary evidence has suggested that cannabidiol (CBD), the non-intoxicating cannabinoid found in cannabis, may mitigate the negative side effects of caffeine (e.g., feeling jittery) without impacting positive or desired effects. CBD also shows potential in reducing undesirable acute effects (e.g., anxiety) of delta-9-tetrahydrocannabinol (THC), the primary intoxicating cannabinoid found in cannabis. Despite these promising findings, little is known about the potential effects of THC, caffeine, and CBD in combination. This double-blind, randomized, placebo-controlled, within-subject crossover study will assess the effects of combinations of THC, CBD, and caffeine (i.e., THC only; THC + caffeine; THC + CBD + caffeine) on subjective energy, arousal, and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Person is between 18 and 55-years-old (inclusive).
2. Person has a body mass index (BMI) between 18 and 35 Kg/m^2 (inclusive).
3. Person is willing and able to provide informed consent.
4. Person has consumed cannabis products containing THC in the past.
5. Person has consumed caffeine products in the past.
6. If person uses medication that has been deemed acceptable (e.g., not contraindicated) by the Investigator, the person has maintained a stable dose and regimen on existing medications for at least 30 days prior to participation in the study and throughout the study.
7. Person agrees to abide by all study restrictions and comply with all study procedures.

Exclusion Criteria:

1. Person has a known history of significant allergic condition or significant hypersensitivity to cannabis, cannabinoid medications, hemp products, or excipients of the investigational product.
2. Person has a known history of significant allergic condition or significant hypersensitivity to caffeine or caffeine products.
3. Person has been exposed to any investigational drug or device < 30 days prior to randomization or plans to take an investigational drug during the study.
4. Person has used cannabis, cannabinoid analogue (e.g., dronabinol, nabilone), and/or any CBD- or delta-9-tetrahydrocannabinol (THC)-containing product within 30 days of screening or during the study.
5. Person has history of use of any synthetic cannabinoid receptor agonist (e.g., spice, K2) within the past year.
6. Person consumes more than 400 mg/day of coffee or other caffeine products (approximately 4 cups of coffee per day) on average within 30 days of screening.
7. Person has used illicit substances (e.g., amphetamine, cocaine, methamphetamine, 3,4-Methyl enedioxy methamphetamine [MDMA], lysergic acid diethylamide [LSD], ketamine, heroin, psilocybin, salvia, prescription medications not prescribed to the person) within 30 days of screening or during the study.
8. Person tests positive for any substance, including THC, at screening.
9. Person is currently using products or medications that may interact with one or more of the ingredients in the investigational product, including the following drugs or supplements: warfarin, clobazam, valproic acid, phenobarbital, mechanistic target of rapamycin [mTOR] inhibitors, oral tacrolimus, St. John's wort, Epidiolex, over the counter stimulants (e.g., phentermine), prescribed stimulants (e.g., Ritalin, Vyvanse), antihypertensive drugs (e.g., captopril, valsartan).
10. Person endorses current suicidal intent as indexed via items 4 and 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS).
11. Person has a history or family history of psychosis or schizophrenia.
12. Person has a diagnosis of cardiac disease or significant cardiac condition.
13. Person has a diagnosis of hypertension and/or a blood pressure reading with systolic pressure > 150 mm Hg or diastolic pressure > 90 mm Hg.
14. Person has an acute or progressive disease or disorder that is likely to interfere with the objectives of the study or the ability to adhere to protocol requirements.
15. Person is currently pregnant, breastfeeding, or is planning to become pregnant within 30 days of completing the study.
16. Woman of childbearing potential, unless she has not engaged in vaginal intercourse, or she has used effective contraception when doing so (for example, double barrier), for at least 30 days prior to the study (however, a male condom should not be used in conjunction with a female condom).
17. Woman of childbearing potential, unless willing to ensure that she or her partner use effective contraception (for example, double barrier) during the study and for 30 days thereafter (however, a male condom should not be used in conjunction with a female condom).
18. Man whose partner is of childbearing potential, unless willing to ensure that he or his partner use effective contraception (for example, double barrier) during the study and for 30 days thereafter (however, a male condom should not be used in conjunction with a female condom).
19. Person has history of diagnosis related to hepatic function and/or significantly impaired hepatic function (alanine aminotransferase [ALT] >5 ⋅ upper limit of normal or total bilirubin [TBL] >2 ⋅ upper limit of normal) OR the ALT or aspartate aminotransferase (AST) >3 ⋅ upper limit of normal and TBL >2 ⋅ upper limit of normal (or international normalized ratio [INR] >1.5).
20. Person demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Change in Driving Performance on the DRiving Under the Influence of Drugs (DRUID®) | 0-, 30-, 90-, 150-, 170-, 240-, 360-, and 480- minutes post drug administration
  Driving Performance as Measured by the DRiving Under the Influence of Drugs (DRUID®) behavioral task. Higher scores = greater impairment.
Driving Performance on the Driving Simulator | 170-minutes post drug administration
  Driving Performance as Measured by a Driving Simulator task

SECONDARY OUTCOMES:
Change in subjective feelings of energy | 0-, 30-, 90-, 150-minutes post drug administration
  Ratings on the Energetic vs. Lethargic item on the Visual Analogue Mood Scale (VAMS)
Change in subjective feelings of alertness | 0-, 30-, 90-, 150-minutes post drug administration
  Ratings on the Alertness vs. Drowsy item on the Visual Analogue Mood Scale (VAMS)
Change in subjective feelings of focus | 0-, 30-, 90-, 150-minutes post drug administration
  Ratings on the Attentive vs. Dreamy item on the Visual Analogue Mood Scale (VAMS)
Change in subjective feelings of jitteriness | 0-, 30-, 90-, 150-minutes post drug administration
  Ratings on the jitteriness item on the Mood Rating Scale (MRS)
Change in subjective feelings of anxiety | 0-, 30-, 90-, 150-minutes post drug administration
  Ratings on the state version of the State-Trait Anxiety Inventory (STAI-S)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Strickland, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine BPRU, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No